CLINICAL TRIAL: NCT05341440
Title: Deciphering the Salutogenic Effects of Close Relationships: Psycho-physiological Coregulation Processes and Their Outcomes in Couples Coping With Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Noa Vilchinsky, prof., Bar-Ilan University, Israel
Other Study IDs: 27122021
Record Dates: First submitted 2022-03-28; First posted 2022-04-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The established attachment theory elucidates how early human bonds bring about functional neurophysiological alterations influencing the lifelong capacity for self and co- regulation within relationships. Based on this framework, the study will investigate potential psycho-physiological co-regulation processes in couples coping with cardiovascular disease, which may explain the established link between relationship satisfaction and recovery outcomes. In the proposed prospective, longitudinal study, the investigators will follow 81 volunteer couples in which one member has experienced an Acute Coronary Syndrome and assess their levels of interactive behavioral synchrony and the accompanying physiological synchrony (the mutual coordination of spouses' autonomic nervous systems), and stress buffering (reduced reactivity to stress in the individual) as assessed by Heart Rate Variability, and Galvanic Skin Response. It is hypothesized that higher levels of physiological synchrony and stress buffering will be associated with enhanced behavioral synchrony in the lab as well as patient outcomes three months later, on three dimensions: emotional (anxiety and depression reduction); behavioral (smoking cessation, medication adherence, cardiac rehabilitation participation) and physical (weight reduction, increased fitness).

ELIGIBILITY:
Inclusion Criteria:

* First Acute Coronary Syndrome
* In a committed relationship lasting over a year
* Registration at the Cardiac Prevention and Rehabiliation Center (CPRC)

Exclusion Criteria:

* A history of previous cardiac events
* A diagnosis other than Acute Coronary Syndrome, co-morbid conditions (such as cancer),
* Lack of Hebrew as a native language.
* Exclusion criteria for partners will be severe co-morbid conditions with life expectancy of less than 6 months (such as advanced cancer) and lack of Hebrew as a native language.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will be male patients with the diagnosis of a first Acute Coronary Syndrome who have been registered in the cardiac prevention and rehabilitation center (CPRC) and are in a committed relationship (i.e., cohabiting for at least one year).
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-03-22 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 3 months
  contains 14 items and consists of two subscales: anxiety and depression. Each item is rated on a four-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represents 'borderline' and 0-7 'normal'.
The Warwich-Edinburgh Mental Well-being Scale | 3 months
  A scale of 14 positively worded items for assessing a population's mental wellbeing. Scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.
Smoking cessation | 3 months
  Smoking cessation will be defined as the delta between the number of cigarettes smoked before the cardiac event and the number of cigarettes smoked 3 months after the start of rehabilitation.
The Medication Adherence Report Scale | 3 months
  Patients will be asked to report on their medication adherence, using the Medication Adherence Rating Scale. Responses are summed for a total score ranging between 5 and 25, with higher scores indicating a higher level of adherence.
Cardiac rehabilitation participation | 3 months
  The number of times patients participated in supervised exercise in the Cardiac Rehabilitation Center. Information regarding Rehabilitation participation will be retrieved from patients' computerized entry files.
Weight change | 3 months
  Weight change is defined as the delta between patients' body-mass index (BMI) from the beginning of rehabilitation and 3 months in.
Fitness change | 3 months
  Will be defined as the change in delta between 3 months after the start of rehabilitation ergometry score and the start of rehabilitation ergometry score (in Metabolic Equivalent of Task Score- METs).

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Hamercaz, Israel